CLINICAL TRIAL: NCT01268592
Title: Vitrification of Oocytes From Female Cancer Patients to Preserve Their Fertility Potential
Brief Title: Fertility Preservation in Female Cancer Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study technique has been declared part of standard care
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10-204A
Record Dates: First submitted 2010-11-01; First posted 2010-12-31 (Estimated); Last update posted 2013-04-23 (Estimated); Status verified 2013-04

CONDITIONS: Fertility
Keywords: fertility preservation; oocyte cryopreservation; vitrification; egg freezing; fertility preservation in female cancer patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- positive cancer diagnosis (Experimental): female patients diagnosed with cancer who wish to preserve their fertility by vitrifying their oocytes
  Interventions: Procedure: oocyte vitrification

INTERVENTIONS:
Procedure: oocyte vitrification — freezing of the patient's retrieved oocytes via vitrification (rapid freezing)

SUMMARY:
The purpose of this study is to preserve the fertility potential in females diagnosed with cancer by vitrifying (rapidly freezing) their oocytes (eggs) before undergoing treatment for their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 14-42 year old females with a cancer diagnosis.
* Clearance letter from treating oncologist.
* Approval by program oncologist or her designee.
* Informed consent has to be signed after consultation with the program physician. Minors require consent of a parent or a legal guardian and assent from the participant.
* Life expectancy (predicted by their malignancy) of 5 or more years.
* Cancer diagnosis should have an expected cure rate of 50% or more, based upon clinico-pathologic features.

Exclusion Criteria:

* Patients whose oncologist and the program oncologist concur that immediate oncologic care should be rendered, not allowing sufficient time for a course of gonadotropin therapy and egg retrieval.
* FSH level >20 MIU/ml, indicating abnormal ovarian function.
* Patients with stage IV cancers (*age appropriate women with stage IV advanced Hodgkin's Lymphoma will be considered, as there is a significant long term survival rate with this advanced disease).
* Patients with incurable cancer diagnoses.
* Patients who are unable or unwilling to sign the informed consent.
* Women cannot have an embryo transfer beyond age 50.

Ages: 14 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2010-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
successful pregnancy | nine months after transfer of embryo(s)
  the primary objective of this study is the establishment of a successful pregnancy, following a disease-free interval after treatment for her cancer; this interval will be patient-dependent and will undoubtedly vary between participants.

SECONDARY OUTCOMES:
impact of stimulation on cancer recurrence | 5 years after treatment
  patients will be followed for five years following cancer treatment to assess the risks associated with ovarian stimulation and the recurrence of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Avner Hershlag, MD, Principal Investigator — Center for Human Reproduction
Locations (1):
- Center for Human Reproduction, Manhasset, New York, United States

REFERENCES:
- [Background] Ajala T, Rafi J, Larsen-Disney P, Howell R. Fertility preservation for cancer patients: a review. Obstet Gynecol Int. 2010;2010:160386. doi: 10.1155/2010/160386. Epub 2010 Mar 31. PMID 20379357
- [Background] Azim AA, Costantini-Ferrando M, Oktay K. Safety of fertility preservation by ovarian stimulation with letrozole and gonadotropins in patients with breast cancer: a prospective controlled study. J Clin Oncol. 2008 Jun 1;26(16):2630-5. doi: 10.1200/JCO.2007.14.8700. PMID 18509175
- [Background] Azim AA, Costantini-Ferrando M, Lostritto K, Oktay K. Relative potencies of anastrozole and letrozole to suppress estradiol in breast cancer patients undergoing ovarian stimulation before in vitro fertilization. J Clin Endocrinol Metab. 2007 Jun;92(6):2197-200. doi: 10.1210/jc.2007-0247. Epub 2007 Mar 13. PMID 17356042
- [Background] Blatt J. Pregnancy outcome in long-term survivors of childhood cancer. Med Pediatr Oncol. 1999 Jul;33(1):29-33. doi: 10.1002/(sici)1096-911x(199907)33:13.0.co;2-2. PMID 10401494
- [Background] Ethics Committee of the American Society for Reproductive Medicine. Fertility preservation and reproduction in cancer patients. Fertil Steril. 2005 Jun;83(6):1622-8. doi: 10.1016/j.fertnstert.2005.03.013. PMID 15950628
- [Background] Ganz PA. Breast cancer, menopause, and long-term survivorship: critical issues for the 21st century. Am J Med. 2005 Dec 19;118 Suppl 12B:136-41. doi: 10.1016/j.amjmed.2005.09.047. PMID 16414339
- [Background] Gook DA, Edgar DH. Human oocyte cryopreservation. Hum Reprod Update. 2007 Nov-Dec;13(6):591-605. doi: 10.1093/humupd/dmm028. Epub 2007 Sep 10. PMID 17846105
- [Background] Grifo JA, Noyes N. Delivery rate using cryopreserved oocytes is comparable to conventional in vitro fertilization using fresh oocytes: potential fertility preservation for female cancer patients. Fertil Steril. 2010 Feb;93(2):391-6. doi: 10.1016/j.fertnstert.2009.02.067. Epub 2009 May 12. PMID 19439285
- [Background] Jeruss JS, Woodruff TK. Preservation of fertility in patients with cancer. N Engl J Med. 2009 Feb 26;360(9):902-11. doi: 10.1056/NEJMra0801454. No abstract available. PMID 19246362
- [Background] Knopman JM, Noyes N, Talebian S, Krey LC, Grifo JA, Licciardi F. Women with cancer undergoing ART for fertility preservation: a cohort study of their response to exogenous gonadotropins. Fertil Steril. 2009 Apr;91(4 Suppl):1476-8. doi: 10.1016/j.fertnstert.2008.07.1727. Epub 2008 Sep 18. PMID 18804204
- [Background] Quintero RB, Helmer A, Huang JQ, Westphal LM. Ovarian stimulation for fertility preservation in patients with cancer. Fertil Steril. 2010 Feb;93(3):865-8. doi: 10.1016/j.fertnstert.2008.10.007. Epub 2008 Nov 14. PMID 19013563
- [Background] Kumayama M and Kato O. All-round vitrification method for human oocytes and embryos. J Asst Reprod Gen 17:447, 2000.
- [Background] Nagy ZP, Chang CC, Bernal DP, Shapiro D, Mitchell-Leef D and Kort HI. Comparison of laboratory and clinical outcomes between fresh and vitrified sibling oocytes obtained from 30-39 year old IVF patients. Fertil Steril 92, Supp3:S67, 2009.
- [Background] Nagy ZP, Chang CC, Shapiro DB, Bernal DP, Elsner CW, Mitchell-Leef D, Toledo AA, Kort HI. Clinical evaluation of the efficiency of an oocyte donation program using egg cryo-banking. Fertil Steril. 2009 Aug;92(2):520-6. doi: 10.1016/j.fertnstert.2008.06.005. Epub 2008 Aug 9. PMID 18692830
- [Background] Noyes N, Boldt J, Nagy ZP. Oocyte cryopreservation: is it time to remove its experimental label? J Assist Reprod Genet. 2010 Feb;27(2-3):69-74. doi: 10.1007/s10815-009-9382-y. Epub 2010 Feb 6. PMID 20140641
- [Background] Oktay K, Hourvitz A, Sahin G, Oktem O, Safro B, Cil A, Bang H. Letrozole reduces estrogen and gonadotropin exposure in women with breast cancer undergoing ovarian stimulation before chemotherapy. J Clin Endocrinol Metab. 2006 Oct;91(10):3885-90. doi: 10.1210/jc.2006-0962. Epub 2006 Aug 1. PMID 16882752
- [Background] Porcu E, Bazzocchi A, Notarangelo L, Paradisi R, Landolfo C, Venturoli S. Human oocyte cryopreservation in infertility and oncology. Curr Opin Endocrinol Diabetes Obes. 2008 Dec;15(6):529-35. doi: 10.1097/MED.0b013e3283199129. PMID 18971682
- [Background] Practice Committees of the American Society for Reproductive Medicine and the Society for Assisted Reproductive Technology. Mature oocyte cryopreservation: a guideline. Fertil Steril. 2013 Jan;99(1):37-43. doi: 10.1016/j.fertnstert.2012.09.028. Epub 2012 Oct 22. PMID 23083924